CLINICAL TRIAL: NCT07274683
Title: Effect of Stellate Ganglion Block on Postoperative Sleep Status in Patients With Prolonged Disorders of Consciousness: a Single--Centre Cohort Study
Brief Title: Stellate Ganglion Block on Postoperative Sleep Status in Patients With Prolonged Disorders of Consciousness
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director, Beijing Tiantan Hospital
Other Study IDs: LJH20250928
Record Dates: First submitted 2025-11-15; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-09

CONDITIONS: Stellate Ganglion Block; Prolonged Disorders of Consciousness; Sleep
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stellate ganglion block: preoperative administration of stellate ganglion block
  Interventions: Drug: stellate ganglion block with 0.5% ropivacaine

INTERVENTIONS:
Drug: stellate ganglion block with 0.5% ropivacaine — A single dose of ultrasound-guided stellate ganglion block with 0.5% ropivacaine was administered to the pDoC patients after induction of general anesthesia but before surgical incision.

SUMMARY:
The goal of this clinical trial is to learn about the effect of preoperative administration of stellate ganglion block on postoperative sleep status in patients with prolonged disorders of consciousness. The main aims to answer are: • To explore the effect of preoperative administration of stellate ganglion block on postoperative polysomnography and total sleep time in patients with prolonged disorders of consciousness. • To explore the effect of preoperative administration of stellate ganglion block on postoperative cerebral oxygen saturation, cerebral hemodynamic parameters and recovery of consciousness. Participants will be pDoC patients with intact skulls after acquired brain injury who will undergo spinal cord electronic stimulator implantation under general anesthesia at Beijing Tiantan Hospital. Stellate ganglion block will be administrated before the surgery. Polysomnography, total sleep time, cerebral oxygen saturation, cerebral hemodynamic parameters, CRS-R scores, GCS scores, WHIM scores and NCS scores will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years;
* Prolonged disorders of consciousness after acquired brain injury;
* Scheduled to undergo spinal cord electronic stimulator implantation under general anesthesia;
* The skull is intact;
* Informed consent is obtained;

Exclusion Criteria:

* Continuous sedation therapy is performed within 72 hours prior to the study;
* The integrity of brain structure is disrupted due to causes such as open head injury and cerebral parenchymal resection;
* Decreased intracranial compliance caused by hydrocephalus and other reasons;
* Airway stenosis or severe dysfunction of ventilation or gas exchange due to various causes;
* Known or suspected severe cardiac, pulmonary, and renal dysfunction;
* History of sedative drug allergy;
* Complicated by other mental or neurological disorders;
* Local anesthetic allergy;
* Other reasons for ineligibility in this study;
* Informed consent is not obtained;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pDOC Patients from Beijing Tian Tan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | on the first postoperative night
  total sleep time on PSG

SECONDARY OUTCOMES:
cerebral oxygen saturation | 30 minutes after stellate ganglion block
  Regional cerebral oxygen saturation (rSO₂) measured by near-infrared spectroscopy (NIRS).
cerebral hemodynamic parameters | 30 minutes after stellate ganglion block.
  cerebral hemodynamic parameters measured by Transcranial Doppler（TCD）
the recovery of consciousness | 1 and 30 days postoperatively
  Consciousness recovery will be assessed using the Coma Recovery Scale-Revised (CRS-R). It assesses patients across six functional domains: auditory, visual, motor, oromotor/verbal, communication, and arousal. The total score ranges from 0 to 23, with higher scores indicating a higher level of consciousness.
Length of ICU stay | 30 days postoperatively
Costs of ICU stay | 30 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tian Tan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
All data generated or analysed during this study will be included in published article. The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: The data that support the findings of this study are available from the corresponding author upon reasonable request.